CLINICAL TRIAL: NCT06028061
Title: Evaluation of The Postoperative Analgesic Effectivity of Quadratus Lumborum Block III With Adjuvant on Patients Undergoing Laparoscopic Cholecystectomy Surgery : A Randomised Controled Study
Brief Title: Evaluation of Effectivity of Quadratus Lumborum Blocks With Adjuvant
Acronym: AdjuvantQLB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, SERPİL ŞEHİRLİOĞLU, MD, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GaziosmanpasaTREHBB
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Pain Management; Postoperative Pain; Analgesia; Nerve Blocks; Nerve Block Duration; Cholecystectomy
Keywords: postoperative pain; laparoscopic cholecystectomy; quadratus lumborum block; abdominal wall blocks; adjuvant; dexamethasone; postoperative analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Adjuvants, Pharmaceutic; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant-free Quadratus lumborum block (Active Comparator): Patients are placed in the lateral decubitus position. The area where the block will be applied is disinfected with povidine iodine. A convex ultrasound probe is placed on the midaxillary line above the iliac crest. By visualizing the transverse process adjacent to the psoas major and quadratus lumborum muscles, using the in-plane technique, using a 22 gauge 80 mm peripheral block needle after negative aspiration into the anterior layer of the thoracolumbar fascia anterior to the quadratus lumborum muscle muscle, 0.5-1 ml of serum After observing hydrodissection with physiological, 20 ml of 0.25% bupivacaine is injected. The same is done to the opposite side.
  Interventions: Procedure: Adjuvant-free Quadratus lumborum block
- Quadratus Lumborum Block with adjuvant (Active Comparator): The same block was applied to this group, but a different local anesthetic mixture was used. Patients are placed in the lateral decubitus position. The area where the block will be applied is disinfected with povidine iodine. A convex ultrasound probe is placed on the midaxillary line above the iliac crest. By visualizing the transverse process adjacent to the psoas major and quadratus lumborum muscles, using the in-plane technique, using a 22 gauge 80 mm peripheral block needle after negative aspiration into the anterior layer of the thoracolumbar fascia anterior to the quadratus lumborum muscle muscle, 0.5-1 ml of serum After observing hydrodissection with physiological, 20 ml of 0.25% bupivacaine and 4mg dexamethasone is injected. The same is done to the opposite side.
  Interventions: Procedure: Quadratus lumborum block III with Adjuvant

INTERVENTIONS:
Procedure: Adjuvant-free Quadratus lumborum block — Patients are placed in the lateral decubitus position. The area where the block will be applied is disinfected with povidine iodine. A convex ultrasound probe is placed on the midaxillary line above the iliac crest. By visualizing the transverse process adjacent to the psoas major and quadratus lumborum muscles, using the in-plane technique, using a 22 gauge 80 mm peripheral block needle after negative aspiration into the anterior layer of the thoracolumbar fascia anterior to the quadratus lumborum muscle muscle, 0.5-1 ml of serum After observing hydrodissection with physiological, 20 ml of 0.25% bupivacaine is injected. The same is done to the opposite side.
  Other Names: only bupivacain, adjuvan-free
  Arms: Adjuvant-free Quadratus lumborum block
Procedure: Quadratus lumborum block III with Adjuvant — The same block was applied to this group too, but a different local anesthetic mixture was used.Patients are placed in the lateral decubitus position. The area where the block will be applied is disinfected with povidine iodine. A convex ultrasound probe is placed on the midaxillary line above the iliac crest. By visualizing the transverse process adjacent to the psoas major and quadratus lumborum muscles, using the in-plane technique, using a 22 gauge 80 mm peripheral block needle after negative aspiration into the anterior layer of the thoracolumbar fascia anterior to the quadratus lumborum muscle muscle, 0.5-1 ml of serum After observing hydrodissection with physiological, 20 ml of 0.25% bupivacaine and 4mg dexamethasone is injected. The same is done to the opposite side.
  Other Names: bupivacain with dexamethasone
  Arms: Quadratus Lumborum Block with adjuvant

SUMMARY:
İn recent years abdominal wall blocks are widely used for to reduce intraoperative anesthetic recuirements and postoperative analgesia.Quadratus lumborum blocks are one of the abdominal wall blocks to used at laparoscopic cholecystectomy.Conventionally adjuvants used to improve and prolonged the effect of periferic nerve, spinal and abdominal blocks.İn this study investigators will evaluate the effectiveness of adjuvants at quatratus lumborum block at patient underwent laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Laparoscopic approach in cholecystectomy surgery is frequently preferred because of its advantages in systemic complications, morbidity, mortality and hospital stay. Pain is one of the important causes of late discharge after surgery. Laparoscopic cholecystectomy surgery requires a multimodal analgesia approach because of its multiple pain components.Regional analgesia techniques are effective in reducing the side effects such as intraoperative opioid use, postoperative pain and nausea and vomiting. Quadratus lumborum III block is a regional technique performed for multimodal analgesia.Adjuvants are known to improve the analgesic efficacy and prolonge the effect of the periferic and central nerve blocks.The aim of this study is to determine the effectiveness of adding adjuvant at quadratus lumborum block for patients who underwent laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria: American Society of Anesthesiologists physical statusⅠ-II

Exclusion Criteria:

* Inclusion Criteria:
* 18-65 years of age
* American Society of Anesthesiologists physical statusⅠ-II

Exclusion Criteria:

* local anesthetic allergy
* Infection at the procedure site Body Mass Index >35 kg/m2 Anticoagulant use with bleeding disorder Chronic analgesia and opioid use with mental and psychiatric disorders Contraindications to regional anesthesia several lung and heart disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Total amount of opioid requirements | within 24 hours after the surgery
  The total tramadol use of the patients in 24 hours will be recorded.
rescue analgesia | within 24 hours after the surgery
  The rescue analgesia requirement and time of the need of the rescue analgesia requirement

SECONDARY OUTCOMES:
intraoperative remifentanil consumption | during operation procedure]
  The total remifentanil use to be used in the maintenance of 0.05-0.2 mcg/kg remifentanil will be recorded by titration according to the hemodynamic data of the intraoperative patients.
Visual Analogue Scale values | at 1st, 4th,8th 12th and 24th hours after the surgery]
  Visual Analogue Scale is a scale of 0-10 cm in length, expressed by non-standard verbal descriptors (no pain-unbearable pain..) indicating the limits of pain intensity on both sides, horizontally or vertically.
side effects such as nausea, vomiting and shoulder pain | within 24 hours after the surgery
  The incidence of postoperative side effects such as nausea, vomiting and shoulder pain will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: SERPİL SEHİRLİOGLU, MD, Principal Investigator — Gaziosmanpasa Research and Education Hospital; BATUHAN BURHAN, MD, Principal Investigator — Gaziosmanpasa Research and Education Hospital; DONDU GENC MORALAR, MD, Study Director — Gaziosmanpasa Research and Education Hospital
Locations (1):
- Gaziosmanpasa Research and Education Hospital, Istanbul, Marmara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Y, Wang YP, Wang HT, Xu YC, Lv HM, Yu Y, Wang P, Pei XD, Zhao JW, Nan ZH, Yang JJ. Ultrasound-guided quadratus lumborum block provided more effective analgesia for children undergoing lower abdominal laparoscopic surgery: a randomized clinical trial. Surg Endosc. 2022 Dec;36(12):9046-9053. doi: 10.1007/s00464-022-09370-z. Epub 2022 Jun 28. PMID 35764836
- [Background] Aygun H, Kavrut Ozturk N, Pamukcu AS, Inal A, Kiziloglu I, Thomas DT, Tulgar S, Nart A. Comparison of ultrasound guided Erector Spinae Plane Block and quadratus lumborum block for postoperative analgesia in laparoscopic cholecystectomy patients; a prospective randomized study. J Clin Anesth. 2020 Jun;62:109696. doi: 10.1016/j.jclinane.2019.109696. Epub 2019 Dec 18. PMID 31862217
- [Background] Herman JA, Urits I, Kaye AD, Urman RD, Viswanath O. Erector Spinae Plane Block (ESPB) or Quadratus Lumborum Block (QLB-II) for laparoscopic cholecystectomy: Impact on postoperative analgesia. J Clin Anesth. 2020 Nov;66:109958. doi: 10.1016/j.jclinane.2020.109958. Epub 2020 Jun 17. No abstract available. PMID 32563073
- [Background] Arafa SK, Elsayed AA, Hagras AM, Shama AAA. Pediatric Postoperative Pain Control With Quadratus Lumborum Block and Dexamethasone in Two Routes With Bupivacaine: A Prospective Randomized Controlled Clinical Trial. Pain Physician. 2022 Oct;25(7):E987-E998. PMID 36288584